CLINICAL TRIAL: NCT05113407
Title: Observatory on the Use of the Shockwave Medical C2 Coronary Lithotripsy System in the General Population in France.
Acronym: France LILI
Status: Recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01876-35
Record Dates: First submitted 2021-10-14; First posted 2021-11-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Lithotripsy; Angioplasty; Coronary Balloon
Keywords: Lithotripsy; Coronary calcified lesion; coronary angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary angioplasty performed using the Shockwave Medical C2 Coronary Lithotripsy System

SUMMARY:
Coronary calcified lesions will have an increasing impact in the daily practice of coronary angioplasty, considering the epidemiological explosion of factors favoring coronary calcifications, first of all diabetes. Moreover, calcified lesions are underestimated in angiography and associated with an increase in angiographic complications, as well as with a worse clinical prognosis. The usual techniques for the preparation of calcified plaque, in particular rotary atherectomy, have a low penetration rate in France (3% of procedures) and are associated with an increase in per-procedural complications without clinical evidence of effectiveness4. A new device has been developed by Schockwave Medical Inc. for the treatment of calcified lesions to facilitate stent delivery: the C2 Shockwave Medical® Coronary Lithotripsy System (IVL), Inc. This system uses the principle of lithotripsy to induce microfractures in the calcified plaque prior to low-pressure balloon dilatation. The objective of the study is to evaluate the safety and performance of the C2 Shockwave Medical® (IVL), Inc. coronary lithotripsy system in coronary angioplasty in the general population in France.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient affiliated to the National Health Insurance System
* Patient for whom a coronary angioplasty procedure is performed using the Shockwave Medical C2 Coronary Lithotripsy System
* For indications of stent malexpansions, stent malexpansion must be defined by: a) angiography: stent malexpansion >30% (QCA and/or stent magnification) b) endocoronary OCT/IVUS imaging with MSA (Minimal Stent Area) <4.5 mm2 or a ratio of MSA/MLA on reference segment<0.8
* Patient willing to participate in the registry

Exclusion Criteria:

* Patient under 18 years of age
* Pregnant or breastfeeding patient
* Patient refusing to participate in the study or unable to give informed consent (patient under guardianship, curatorship or legal guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included in cardiology departments participating in the study. The study may be offered to any patient undergoing coronary artery angioplasty using the Shockwave Medical C2 coronary lithotripsy system.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and performance of the Shockwave Medical® C2 Coronary Lithotripsy System (IVL), Inc. in coronary angioplasty in "all patients" in France. | 1 year after procedure
  Target Vessel Failure (TVF) composite endpoint at 1 year:
  * Cardiac death
  * Myocardial infarction according to ARC II definition of myocardial infarction (unless the infarction is clearly attributable to a non-target vessel)
  * Target vessel revascularization (TVR)

SECONDARY OUTCOMES:
To evaluate the device success | During initial hospitalization, within 2-4 days after procedure
  Ability to deliver the Shockwave Medical Coronary C2 Lithotripsy System to the lesion site to be treated and achieve a residual lesion < 50% after application of acoustic therapy.
To evaluate the procedural success in de novo lesions | During initial hospitalization, within 2-4 days after procedure
  Procedural success is defined as stent placement with < 20% residual stenosis and no serious angiographic complications (i.e., acute dissection (types D through F), perforation, acute obstruction, persistent slow flow or "no reflow").
To evaluate the procedural success in stent malexpansion | During initial hospitalization, within 2-4 days after procedure
  Post-IVL procedural success is defined by a) malexpansion < 20% (QCA and/or Stent magnification) and/or b) endocoronary OCT/IVUS imaging with a MSA (Minimal Stent Area) >4.5 mm2
To evaluate the rate of MACE during the year of follow-up | 1 year after procedure
  Evaluate the rate of events considered as Major adverse cardiac events (MACE classification) : all-cause death, myocardial infarction (including non-target vessel MI), any coronary revascularization.
To evaluate the rate of stent thrombosis during the year of follow-up | 1 year after procedure
  Rate of Stent thrombosis
To evaluate the rate of target lesion failure during the year of follow-up | 1 year after procedure
  Evaluate the rate of Target lesion failure (Device-oriented endpoint) = addition of rates of events like cardiac death, myocardial infarction (unless clearly attributable to a vessel other than the target vessel) and target lesion revascularization (TLR)
To evaluate the rate of per-procedural coronary complications | During initial hospitalization, within 2-4 days after procedure
  Rate of Coronary complication as Dissection (A-F), Slow Flow, No reFlow and abrupt vessel occlusion, Perforation

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin HONTON, Principal Investigator — Clinique Pasteur - France
Locations (1):
- Clinique Pasteur, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee MS, Shah N. The Impact and Pathophysiologic Consequences of Coronary Artery Calcium Deposition in Percutaneous Coronary Interventions. J Invasive Cardiol. 2016 Apr;28(4):160-7. Epub 2015 Aug 25. PMID 26301561
- [Background] Bhatt P, Parikh P, Patel A, Chag M, Chandarana A, Parikh R, Parikh K. Orbital atherectomy system in treating calcified coronary lesions: 3-Year follow-up in first human use study (ORBIT I trial). Cardiovasc Revasc Med. 2014 Jun;15(4):204-8. doi: 10.1016/j.carrev.2014.03.004. Epub 2014 Mar 19. PMID 24746600
- [Background] Genereux P, Madhavan MV, Mintz GS, Maehara A, Palmerini T, Lasalle L, Xu K, McAndrew T, Kirtane A, Lansky AJ, Brener SJ, Mehran R, Stone GW. Ischemic outcomes after coronary intervention of calcified vessels in acute coronary syndromes. Pooled analysis from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) and ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) TRIALS. J Am Coll Cardiol. 2014 May 13;63(18):1845-54. doi: 10.1016/j.jacc.2014.01.034. Epub 2014 Feb 19. PMID 24561145
- [Background] Abdel-Wahab M, Richardt G, Joachim Buttner H, Toelg R, Geist V, Meinertz T, Schofer J, King L, Neumann FJ, Khattab AA. High-speed rotational atherectomy before paclitaxel-eluting stent implantation in complex calcified coronary lesions: the randomized ROTAXUS (Rotational Atherectomy Prior to Taxus Stent Treatment for Complex Native Coronary Artery Disease) trial. JACC Cardiovasc Interv. 2013 Jan;6(1):10-9. doi: 10.1016/j.jcin.2012.07.017. Epub 2012 Dec 19. PMID 23266232
- [Background] Brinton TJ, Ali ZA, Hill JM, Meredith IT, Maehara A, Illindala U, Lansky A, Gotberg M, Van Mieghem NM, Whitbourn R, Fajadet J, Di Mario C. Feasibility of Shockwave Coronary Intravascular Lithotripsy for the Treatment of Calcified Coronary Stenoses. Circulation. 2019 Feb 5;139(6):834-836. doi: 10.1161/CIRCULATIONAHA.118.036531. No abstract available. PMID 30715944
- [Background] Ali ZA, Brinton TJ, Hill JM, Maehara A, Matsumura M, Karimi Galougahi K, Illindala U, Gotberg M, Whitbourn R, Van Mieghem N, Meredith IT, Di Mario C, Fajadet J. Optical Coherence Tomography Characterization of Coronary Lithoplasty for Treatment of Calcified Lesions: First Description. JACC Cardiovasc Imaging. 2017 Aug;10(8):897-906. doi: 10.1016/j.jcmg.2017.05.012. PMID 28797412
- [Background] Ali ZA, Nef H, Escaned J, Werner N, Banning AP, Hill JM, De Bruyne B, Montorfano M, Lefevre T, Stone GW, Crowley A, Matsumura M, Maehara A, Lansky AJ, Fajadet J, Di Mario C. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Stenoses: The Disrupt CAD II Study. Circ Cardiovasc Interv. 2019 Oct;12(10):e008434. doi: 10.1161/CIRCINTERVENTIONS.119.008434. Epub 2019 Sep 25. PMID 31553205
- [Background] Hill JM, Kereiakes DJ, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease. J Am Coll Cardiol. 2020 Dec 1;76(22):2635-2646. doi: 10.1016/j.jacc.2020.09.603. Epub 2020 Oct 15. PMID 33069849
- [Background] Brodmann M, Werner M, Holden A, Tepe G, Scheinert D, Schwindt A, Wolf F, Jaff M, Lansky A, Zeller T. Primary outcomes and mechanism of action of intravascular lithotripsy in calcified, femoropopliteal lesions: Results of Disrupt PAD II. Catheter Cardiovasc Interv. 2019 Feb 1;93(2):335-342. doi: 10.1002/ccd.27943. Epub 2018 Nov 25. PMID 30474206
- [Background] Tovar Forero MN, Wilschut J, Van Mieghem NM, Daemen J. Coronary lithoplasty: a novel treatment for stent underexpansion. Eur Heart J. 2019 Jan 7;40(2):221. doi: 10.1093/eurheartj/ehy593. No abstract available. PMID 30289452
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Derived] Honton B, Benamer H, Cayla G. [France LILI (Intracoronary Lithoplasty)]. Ann Cardiol Angeiol (Paris). 2023 Oct 28;72(6):101692. doi: 10.1016/j.ancard.2023.101692. Online ahead of print. French. PMID 39492363